CLINICAL TRIAL: NCT01821742
Title: Echocardiography in Kids Intensive Care Decision Support - is Focused Echocardiography Superior to Pressure Derived Measurements at Predicting Fluid Responsiveness in Critically Ill Children?
Brief Title: Echocardiography in Kids Intensive Care Decision Support
Acronym: ECHOKIDS
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS ID 121440
Record Dates: First submitted 2013-03-22; First posted 2013-04-01 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Fluid Responsiveness; Cardiac Output
Keywords: Shock; Fluid bolus; Cardiac output; Children in intensive care
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children requiring fluid bolus on PICU
  Interventions: Other: Ultrasound cardiac output measurement

INTERVENTIONS:
Other: Ultrasound cardiac output measurement

SUMMARY:
A study to determine if echocardiographically derived parameters, plethysmographic variability index and pulse pressure variation predict fluid responsiveness in children on PICU.

DETAILED DESCRIPTION:
A study to determine if echocardiographically derived parameters, plethysmographic variability index and pulse pressure variation predict fluid responsiveness in children on PICU. These parameters will be measured pre and post fluid bolus in children prescribed fluid bolus therapy for clinical indications on the PICU. Children will be classified as responders (>10% increase in cardiac output) and non responders (<10% increase). Appropriate statistical tests will be performed to determine the most useful predictor of an increase in cardiac output following a fluid bolus.

ELIGIBILITY:
Inclusion Criteria:

* Any ventilated child requiring fluid bolus therapy on the PICU for clinical indications

Exclusion Criteria:

* Arrythmia
* Intracardiac shunt

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Shocked children on PICU
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Fluid responsiveness | Immediate
  10% increase in cardiac output following fluid bolus

CONTACTS AND LOCATIONS:
Overall Officials: David Inwald, MB BChir, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

REFERENCES:
- [Result] McLean JRL, Inwald DP. The utility of stroke volume variability as a predictor of fluid responsiveness in critically ill children: a pilot study. Intensive Care Med. 2014 Feb;40(2):288-289. doi: 10.1007/s00134-013-3171-x. Epub 2013 Dec 5. No abstract available. PMID 24306083